CLINICAL TRIAL: NCT05441423
Title: Accuracy and Reliability of Ultra Low Dose CBCT Versus CBCT Imaging in Semi-automated Segmentation of the Mandibular Condyle (A Diagnostic Accuracy Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marina Salib, PhD Candidate, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: ORAD7-1-1-1
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: CBCT - Condyle - Semi-automated Segmentation - Ultra-low Dose

STUDY DESIGN:
Intervention Model Description: Dry human skulls and dry human mandibles will be recruited from Anatomy Department, Faculty of Medicine, Cairo University. Human skulls and mandibles will be recruited according to the following eligibility criteria: inclusion criteria will be mandibles with sound condyles and skulls with sound glenoid fossa. Exclusion criteria will be skulls with fractured glenoid fossa, or glenoid fossa with developmental deformities, mandibles with fractured condylar neck or head, presence of pathological lesions, fracture, Shipping, or developmental deformities in the condyle.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CBCT — CBCT Scans. conventional & ultra low dose

SUMMARY:
The objective of this study will be evaluation of accuracy and reliability of CBCT imaging versus Ultra low dose CBCT imaging in semi-automated mandibular condyle segmentation (linear and volumetric assessment of the condyles), in cases requiring condylar and mandibular reconstruction. Dry human skulls and dry human mandibles will be recruited from Anatomy Department, Faculty of Medicine, Cairo University. The following radiographic examination will be done in Oral and Maxillofacial Radiology Department, Faculty Dentistry, Cairo University. they include Radiographic imaging by CBCT machine & Data acquisition and analysis. then semiautomated segmentation will be performed for the mandibular condyles and then after the assessment will be done as both linear and volumetric for each condyle.

DETAILED DESCRIPTION:
The objective of this study will be evaluation of accuracy and reliability of CBCT imaging versus Ultra low dose CBCT imaging in semi-automated mandibular condyle segmentation (linear and volumetric assessment of the condyles), in cases requiring condylar and mandibular reconstruction. Dry human skulls and dry human mandibles will be recruited from Anatomy Department, Faculty of Medicine, Cairo University. The following radiographic examination will be done in Oral and Maxillofacial Radiology Department, Faculty Dentistry, Cairo University. they include Radiographic imaging by CBCT machine & Data acquisition and analysis. then semiautomated segmentation will be performed for the mandibular condyles and then after the assessment will be done as both linear and volumetric for each condyle.

R (Reference standard): Physical real linear measurements of the condyles will be considered as reference standard, where distances will be measured by digital caliper on the dry human in millimeters as supported by García-Sanz et al. (2017) & (Kim et al., 2020).

Volumetric measurements form the dry human condyles will be considered as reference standard where water displacement method will be used (according to Archimedes' principle), by immersion of the condyle under investigation in a water filled graduated transparent glass container, after being hangered from a L-shaped metal hanger by using a rope, till the complete immersion of the condylar volume (which was demarcated by using the gutta percha points) under the water level, this will provide more standardization. Then, the displaced amount of water, will be observed and then aspirated by a graduated pipette to calculate its volume in cubic millimeters. This technique was supported by García-Sanz et al. (2017).

ELIGIBILITY:
Inclusion Criteria:

1. mandibles with sound condyles
2. skulls with sound glenoid fossa.

Exclusion Criteria:

1. skulls with fractured glenoid fossa,
2. glenoid fossa with developmental deformities,
3. mandibles with fractured condylar neck or head,
4. presence of pathological lesions,
5. fracture,
6. Shipping,
7. developmental deformities in the condyle.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Linear Measurements | 1 year
  Linear assessment will be done by applying the same landmarks on the both segmented condyles (yielded rom Conventional and Ultralow dose CBCT imaging), Distances will be measured on the segmented condyles from the segmentation software in millimeters. The linear distances according to García-Sanz et al. (2017) will be as follows:
  * Line 1: Condylar width measured as the distance between lateral and medial landmarks.
  * Line 2: Condylar length measured as distance between anterior and posterior landmarks.
  * Line 3: Condylar height measured as distance of the perpendicular line traced from superior point to line 1.

SECONDARY OUTCOMES:
Volumetric measurements | 1 year
  Volumetric assessment will be done by calculating both segmented condylar volumes (yielded from Conventional and Ultralow dose CBCT imaging) by the segmentation software in cubic millimeters.

IPD SHARING:
Plan to Share IPD: No